CLINICAL TRIAL: NCT07088679
Title: Efficacy of a Natural Bioactive Gel as an Adjunct to Standard Therapy in the Treatment of Peri-Implantitis: A Randomized Controlled Split-Mouth Clinical Trial
Brief Title: Natural Bioactive Gel for Peri-Implantitis
Acronym: PERISTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SMGEL
Record Dates: First submitted 2025-07-05; First posted 2025-07-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Peri-implantitis; Dental Implants; Non-surgical Periodontal Therapy
Keywords: Peri-implantitis; Dental implants; Bioactive gel; Sterify Gel; Non-surgical therapy; Split-mouth design; Oral biofilm; Mechanical debridement; Randomized controlled trial
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sterify Gel + Non-Surgical Therapy (Experimental): This arm receives standard non-surgical peri-implantitis treatment (mechanical debridement, air-polishing with erythritol and glycine) plus the application of Sterify Gel®, a mucoadhesive hydrogel containing polyvinyl polymers, hydroxytyrosol, magnesium ascorbyl phosphate, and nisin, applied in the peri-implant pocket using a sterile needle.
  Interventions: Drug: Sterify Gel (mucoadhesive bioactive gel); Procedure: Standard Non-Surgical Peri-Implantitis Therapy
- Non-Surgical Therapy Only (Active Comparator): This arm receives standard non-surgical peri-implantitis treatment only, including mechanical debridement with ultrasonic and manual instruments, and air-polishing with erythritol and glycine powders. No adjunctive gel is applied.
  Interventions: Procedure: Standard Non-Surgical Peri-Implantitis Therapy

INTERVENTIONS:
Drug: Sterify Gel (mucoadhesive bioactive gel) — Sterify Gel® is a sterile, ready-to-use mucoadhesive hydrogel formulated with polyvinyl polymers, hydroxytyrosol (a natural antioxidant), magnesium ascorbyl phosphate (a stable vitamin C derivative), and nisin (a naturally occurring antimicrobial peptide). In this study, it is applied into the peri-implant pocket using a 0.6 mm - 23GA sterile needle (Gerhò®) immediately after non-surgical debridement. Application is performed at baseline and at follow-up visits (1, 3, 6, and 9 months). Patients are instructed to avoid rinsing, eating, or using oral hygiene aids at the treated sites for at least 2 hours post-application, and to follow specific hygiene instructions for 48 hours.
  Arms: Sterify Gel + Non-Surgical Therapy
Procedure: Standard Non-Surgical Peri-Implantitis Therapy — Standard therapy consists of supra- and subgingival professional mechanical debridement of peri-implant sites using ultrasonic inserts and manual curettes covered with biocompatible materials (PEEK, teflon, or titanium) to avoid damage to the implant surface. This is followed by air-polishing using erythritol powder (Air-Flow Plus®, EMS; 14 µm) for supragingival biofilm removal and glycine powder (Air-Flow Perio®, EMS; 25 µm) for subgingival polishing. This procedure is repeated at baseline and at 1, 3, 6, and 9 months without the adjunctive use of any topical gel.

SUMMARY:
This study is a randomized controlled clinical trial using a split-mouth design to evaluate the effectiveness of a natural bioactive gel (Sterify Gel®) as an adjunct to standard non-surgical therapy for peri-implantitis. Peri-implantitis is an inflammatory disease that affects the tissues around dental implants and can lead to bone loss and implant failure. The goal of the study is to determine whether the application of Sterify Gel®, which contains polyvinyl polymers, hydroxytyrosol, magnesium ascorbyl phosphate, and nisin, can improve clinical outcomes when used in addition to conventional mechanical debridement and air-polishing.

The trial will include 20 patients, each with at least two implants in different quadrants affected by peri-implantitis. One implant will be treated with standard therapy plus the gel (test site), while the other will receive standard therapy alone (control site). Clinical outcomes will be measured over a 9-month period, including plaque levels, bleeding on probing, probing depth, suppuration, and bone loss. The results will help assess whether this gel enhances the effectiveness of routine non-surgical peri-implantitis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years
* Presence of peri-implantitis involving at least two dental implants located in different quadrants
* Presence of bleeding and/or suppuration on probing
* Increased probing depth (PD) and radiographic bone loss compared to previous examinations
* In the absence of previous clinical data: PD ≥ 6 mm and bone loss ≥ 3 mm apically from the coronal portion of the intraosseous implant area (radiographically assessed)
* Willingness and ability to comply with study protocol and follow-up visits
* Written informed consent provided

Exclusion Criteria:

* Patients with cardiac pacemakers or other implanted electronic devices
* Neurological or psychiatric disorders that may interfere with study participation
* Systemic diseases, metabolic disorders, or autoimmune conditions
* Pregnancy or lactation Current participation in other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in peri-implant Modified Plaque Index (mPI) | At baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3), and 9 months (T4)
  The Modified Plaque Index (mPI) is a semi-quantitative index used to assess the presence and accumulation of bacterial plaque around dental implants. Scores are recorded at six peri-implant sites per implant using a 3-point scale, where 0 indicates no plaque, 1 indicates plaque detectable only with a probe, and 2 indicates plaque visible to the naked eye. For each implant, the mean score is calculated. At the patient level, the percentage of sites with a score greater than or equal to 1 is also calculated. The primary outcome is the change in mPI between baseline and the final follow-up, comparing treated and control sites.

SECONDARY OUTCOMES:
Change in percentage of peri-implant sites with Bleeding on Probing (BoP) | At baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3), and 9 months (T4)
  Bleeding on Probing (BoP) is a binary clinical index used to assess inflammation of peri-implant soft tissues. Six peri-implant sites are evaluated per implant. Each site is scored as 0 if no bleeding occurs within 15 seconds of gentle probing, or 1 if bleeding is present. The percentage of bleeding sites is calculated for each patient. The outcome is the change in the percentage of peri-implant sites with BoP ≥1 over time, comparing test and control sites.
Change in peri-implant Bleeding Score (BS) | At baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3), and 9 months (T4)
  The Bleeding Score (BS) assesses bleeding severity upon probing at six sites per implant. Each site is scored on a 4-point scale: 0 = no bleeding, 1 = isolated bleeding points, 2 = continuous bleeding line along the margin, 3 = profuse bleeding. The outcome is the change in the mean BS and the percentage of sites with BS ≥1 over time, calculated at the patient level.
Change in mean peri-implant Probing Depth (PD) | At baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3), and 9 months (T4)
  Probing Depth (PD) is measured at six sites per implant using a calibrated periodontal probe with light force (≤ 0.25 N). It represents the distance in millimeters from the mucosal margin to the base of the pocket. The outcome is the change in mean PD per implant and the percentage of sites with PD ≥4 mm, calculated at the patient level over time.
Change in percentage of peri-implant sites with Suppuration (Suppuration Index, SI) | At baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3), and 9 months (T4)
  Suppuration Index (SI) evaluates the presence of purulent exudate at four peri-implant sites per implant (mesial, distal, buccal, lingual/palatal). Each site is scored as 0 (no suppuration) or 1 (visible suppuration upon probing). The outcome is the change over time in the percentage of sites with suppuration, calculated at the patient level.
Change in peri-implant implant mobility score | At baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3), and 9 months (T4)
  Implant mobility is assessed manually using two rigid instruments. The score is assigned as follows: 0 = no mobility, 1 = perceptible horizontal mobility on manual testing, 2 = clinically visible horizontal mobility, 3 = horizontal and vertical mobility (indication for implant removal). The outcome is the change in implant mobility score over time, evaluated per implant.
Change in percentage of peri-implant sites with Gingival Bleeding Index (GBI) | At baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3), and 9 months (T4)
  The Gingival Bleeding Index (GBI) assesses marginal gingival inflammation. Four sites per implant (mesial, distal, buccal, lingual/palatal) are gently probed. A score of 1 indicates bleeding within 10-15 seconds; 0 indicates absence of bleeding. The outcome is the change in the percentage of sites with GBI = 1 at the patient level over time.
Change in percentage of peri-implant sites with Marginal Mucosal Conditions (MMC) | At baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3), and 9 months (T4)
  Marginal Mucosal Conditions (MMC) assess visible signs of inflammation (redness, edema, altered contour) at four peri-implant sites. Each site is scored as 0 (healthy mucosa) or 1 (clinical signs of inflammation). The outcome is the change in the percentage of sites with MMC = 1 at the patient level over time.
Change in percentage of peri-implant sites with Mucosal Margin Migration (MMM) | At baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3), and 9 months (T4)
  Mucosal Margin Migration (MMM) assesses the presence of apical migration of the mucosal margin compared to baseline. Four sites per implant are examined visually. A score of 0 indicates no migration; 1 indicates visible apical shift. The outcome is the change in the percentage of sites with MMM = 1 at the patient level over time.
Change in peri-implant Radiographic Bone Loss (RBL) | At baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3), and 9 months (T4)
  Radiographic Bone Loss (RBL) is a quantitative parameter used to assess marginal bone loss around dental implants. Standardized intraoral radiographs are obtained using a Rinn-type centering device. For each implant, the distance in millimeters from the implant shoulder to the first visible bone-to-implant contact is measured both mesially and distally. Bone loss is recorded in absolute millimeters and expressed as a percentage of the total implant length. The outcome is the change in mesial and distal RBL values between timepoints, comparing test and control sites.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.